CLINICAL TRIAL: NCT00950781
Title: Cortisol Levels on Menopausal Vasomotor Symptoms - an Ancillary (Addendum) Study to the "Impact of Traditional Acupuncture on Menopausal Vasomotor Symptoms, Psychological Stress and the Hypothalamic Pituitary Adrenal (HPA) - Sympathetic Nervous System (SNS) Axis: A Randomized, Controlled Trial"
Brief Title: Cortisol Levels on Menopausal Symptoms - Ancillary (Addendum) Study to Protocol 16997
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Noel Bairey Merz, Director, Cedars-Sinai Medical Center
Other Study IDs: IRB# 17569
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Menopause
Keywords: Menopause; Cortisol; ACTH
MeSH Terms: interventions — Adrenocorticotropic Hormone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group: Group
  Interventions: Procedure: ACTH

INTERVENTIONS:
Procedure: ACTH — During the ACTH test an IV will be placed in subjects arms, 25mL of blood will be drawn at -30 minutes and 6mL of blood will be drawn at -15 minutes and 0 minutes respectively. Following, 0.25mg of ACTH will be injected intravenous over 60 seconds, and a final 12mL of blood will be drawn 60 minutes later. That is, a total of 50mL of blood will be drawn to test serum blood hormone levels from the subjects during the ACTH (Hormone) Stimulation Test.

SUMMARY:
This is an ancillary study to Protocol 16997 to examine the stress hormone level in women with menopausal symptoms. This ancillary project will collect additional data from the 45 subjects enrolled in Protocol 16997 (no subjects have enrolled in Protocol 16997 so far). This study protocol differs from the main protocol (16997) because it will include an ACTH (Hormone) Stimulation Test which will assess the functioning of stress response in the subjects at entry and exit.

Subjects will undergo the ACTH test for this ancillary protocol in the morning when they complete 24-hour urine collection for Protocol 16997. The ACTH (Hormone) Stimulation Test will not be done in the main protocol 16997. During the ACTH test an IV will be placed in subjects arms, 25mL of blood will be drawn at -30 minutes and 6mL of blood will be drawn at -15 minutes and 0 minutes respectively. Following, 0.25mg of ACTH will be injected intravenous over 60 seconds, and a final 12mL of blood will be drawn 60 minutes later. That is, a total of 50mL of blood will be drawn to test serum blood hormone levels from the subjects during the ACTH (Hormone) Stimulation Test.

The 24 hour cortisol data collected in the main protocol 16997 will be used for this study analysis.

When subjects are consented for Protocol 16997, they will also be consented for this ancillary study. In addition to the consent visit, subjects will have two study specific visits (entry and exit) for this ancillary study. The PI will schedule the specific visits for this study to be in conjunction with those scheduled for Protocol 16997.

There is no collaborations with other sites in the ancillary study.

ELIGIBILITY:
Inclusion Criteria:

1. Women with menopausal VMS bothersome enough to warrant treatment;
2. Minimum of 7 hot flashes per day (on average);
3. Age limits: women ages 40-70 who have had at least one missed menstrual cycle or have undergone spontaneous menopause, women of any age who have medically induced menopause, women of any age who have had oophorectomy;
4. Informed written consent;
5. Ability to follow treatment protocols.

Exclusion Criteria:

Exclusion Criteria (cohort)

1. Concomitant illness with reasonable likelihood of limiting survival to less than one year;
2. Current substance abuse (alcohol or drug);
3. Pregnancy known, suspected or planned in next year.

Exclusion Criteria (TA intervention)

1. Other concomitant menopause treatment;
2. Participating in acupuncture treatment or formal psychological stress management program within the last year;
3. Participating in another treatment for VMS, unless willing to stop it 4 weeks in advance of participation;
4. HIV infection, chronic or active hepatitis or other blood-borne illness.

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Menopausal women
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2009-01; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
circulation at baseline and after acute ACTH stimulation | 2 hours

SECONDARY OUTCOMES:
urine collection of menopausal women with VMS pre and post treatment | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: C. Noel Bairey Merz, MD, Study Director — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Women's Heart Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes